CLINICAL TRIAL: NCT04466566
Title: Effect of Genetic Variation in the GLP-1 Receptor on Beta-cell Function During Fasting and Hyperglycemia in Nondiabetic Humans
Brief Title: A Study to Evaluate the Effect of Genetic Variation on Beta-cell Function During Fasting and Hyperglycemia in Nondiabetics
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Adrian Vella (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor-Investigator, Adrian Vella, Principal Investigator, Mayo Clinic
Organization: Mayo Clinic (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 20-003984; R01DK126206 (NIH)
Record Dates: First submitted 2020-06-30; First posted 2020-07-10 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Healthy
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Saline (Placebo Comparator): Saline will be infused during the study
  Interventions: Other: Saline
- Exendin-9,39 (Active Comparator): Exendin-9,39 will be infused during the study
  Interventions: Biological: Exendin-9,39

INTERVENTIONS:
Other: Saline — Saline will serve as the control
  Arms: Saline
Biological: Exendin-9,39 — Exendin-9,39 will block the GLP-1 receptor
  Arms: Exendin-9,39

SUMMARY:
The GLP-1 receptor (GLP1R) gene is found on the beta cells of the pancreas. Its role is in the control of blood sugar level by enhancing insulin secretion from the pancreas after eating a meal. The purpose of this research study to find out how genetic variations in GLP1R alter insulin secretion, in the fasting state and when blood sugars levels are elevated.

ELIGIBILITY:
Inclusion Criteria:

* 40 nondiabetic subjects will be recruited.
* 20 subjects with the AA genotype at rs3765467 and remainder will have the GG genotype.
* Individuals encompassing the age span of 25-65 years.

Exclusion Criteria:

* Individuals under 25 and over 65 years of age.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2022-10-17 (Actual); Primary Completion 2025-09-30 (Actual); Study Completion 2025-12-30 (Actual)

PRIMARY OUTCOMES:
Insulin secretion quantified using the minimal model to generate an index of beta-cell responsivity (Φ) | This will be calculated from the 0-180 minute data of the study

SECONDARY OUTCOMES:
Glucagon secretion measured by immunoassay | This will be averaged over the 0-180 minute data of the study

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Vella, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials